CLINICAL TRIAL: NCT05428696
Title: A Randomized, Double-blind, Placebo-controlled First-in-Human Study of Single and Multiple Doses of ALXN2080 in Healthy Participants
Brief Title: Safety and Tolerability, PK, and PD Study of Single and Multiple ALXN2080 Doses in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALXN2080-HV-101
Record Dates: First submitted 2022-04-26; First posted 2022-06-23 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: ALXN2080; Complement system; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- SAD - Cohort 1 (Experimental): Eight participants will receive a single dose of Dose Amount 1 of ALXN2080, and 2 participants will receive placebo.
  Interventions: Drug: ALXN2080; Drug: Placebo
- SAD - Cohort 2 (Experimental): Eight participants will receive a single dose of Dose Amount 2 of ALXN2080, and 2 participants will receive placebo.
  Interventions: Drug: ALXN2080; Drug: Placebo
- SAD - Cohort 3 (Experimental): Eight participants will receive a single dose of Dose Amount 3 of ALXN2080, and 2 participants will receive placebo.
  Interventions: Drug: ALXN2080; Drug: Placebo
- SAD - Cohort 4 (Experimental): Eight participants will receive a single dose of Dose Amount 4 of ALXN2080, and 2 participants will receive placebo.
  Interventions: Drug: ALXN2080; Drug: Placebo
- SAD - Cohort 5 (Experimental): Eight participants will receive a single dose of Dose Amount 5 of ALXN2080, and 2 participants will receive placebo.
  Interventions: Drug: ALXN2080; Drug: Placebo
- SAD - Cohort 6 (Experimental): Eight participants will receive a single dose of Dose Amount 6 of ALXN2080, and 2 participants will receive placebo.
  Interventions: Drug: ALXN2080; Drug: Placebo
- MAD - Cohort 1 (Experimental): Eight participants will receive multiple doses of Dose Amount A of ALXN2080 at a Dosing Frequency 1, and 2 participants will receive placebo for 14 days.
  Interventions: Drug: ALXN2080; Drug: Placebo
- MAD - Cohort 2 (Experimental): Eight participants will receive multiple doses of Dose Amount B of ALXN2080 at a Dosing Frequency 1, and 2 participants will receive placebo for 14 days.
  Interventions: Drug: ALXN2080; Drug: Placebo
- MAD - Cohort 3 (Experimental): Eight participants will receive multiple doses of Dose Amount C of ALXN2080 at a Dosing Frequency 1 or Frequency 2, and 2 participants will receive placebo for 14 days.
  Interventions: Drug: ALXN2080; Drug: Placebo
- MAD - Cohort 4 (Experimental): Eight participants will receive multiple doses of Dose Amount D of ALXN2080 at a Dosing Frequency 1 or Frequency 2, and 2 participants will receive placebo for 14 days.
  Interventions: Drug: ALXN2080; Drug: Placebo

INTERVENTIONS:
Drug: ALXN2080 — Powder-in-capsule
Drug: Placebo — Powder-in-capsule

SUMMARY:
This study is designed to evaluate the safety and tolerability, pharmacokinetics and pharmacodynamics of single and multiple doses of ALXN2080 in healthy adult participants.

DETAILED DESCRIPTION:
Participants will be assigned to 10 different cohorts (6 SAD cohorts and 4 MAD cohorts), each with 8 participants on active treatment with ALXN2080 and 2 participants on placebo. ALXN2080 will be administered under fasted conditions throughout this study, except for the last SAD Cohort 6 in which ALXN2080 will be given with food to evaluate the effect of food on the single-dose pharmacokinetics of ALXN2080.

ELIGIBILITY:
Inclusion Criteria:

* Healthy is defined as having no clinically relevant abnormalities identified by a detailed medical history, physical examination, blood pressure and heart rate measurements, 12-lead ECG, and clinical laboratory tests.
* Body mass index (BMI) of 18 to 30 kg/m2 with a minimum body weight of 50 kg. BMI max is 32 kg/m2.
* Male or female; female of childbearing potential and male participants agreed to follow protocol specified contraception guidance.

Exclusion Criteria:

* Significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders.
* History of hypersensitivity to any ingredient contained in the study intervention.
* Evidence of active infections, history of meningococcal infection, unexplained, or recurrent infection.
* Known or suspected history of drug or alcohol abuse or dependence.
* Current tobacco users or smokers.
* Diseases or conditions or previous procedures known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* For females: pregnant, breastfeeding, or intending to conceive during the course of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Day 1 through up to Day 28

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve Extrapolated to Infinity (AUC0-inf) Of Single Dose ALXN2080 | Up to 168 hours postdose
Maximum Observed Plasma Concentration (Cmax) of Single Dose ALXN2080 | Up to 168 hours postdose

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.